CLINICAL TRIAL: NCT05193305
Title: Study of Healthy Cohort for Early Detection of Cancer
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00301815
Record Dates: First submitted 2021-12-29; First posted 2022-01-14 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected yearly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cancer produces a significant burden on society with a majority diagnosed at late stages when the chance of cure is low. Early diagnosis improves patient outcomes. Data consisting of lifestyle factors, medications, physical activity, years before conventional cancer diagnosis is also worthwhile for to determine early detection. This is only achievable with longitudinal tracking of a large number of healthy individuals and identifying those who do develop cancer over time.

DETAILED DESCRIPTION:
To conduct a longitudinal cohort study of patients who do not have a malignancy at the time of enrollment and are followed over a 20 year period to see if patients develop a malignancy and associate clinical and lifestyle factors as well as collection of blood. All adults 18 years of age and older undergoing upper or lower endoscopy for routine medical care will be eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

* All adults 18 years of age of older undergoing upper or lower endoscopy for routine medical care.

Exclusion Criteria:

* Persons with current malignancy
* Persons with history of malignancy and treatment within last 5 years of enrollment, excluding non-melanoma skin cancer or cervical in-situ.
* Persons who are unable or unwilling to provide repeat blood samples and complete follow-up questionnaires
* Persons who lack the capacity to provide consent
* Persons who do not speak English
* Persons who are visually or hearing impaired.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Prospective participants who are to undergo upper or lower gastrointestinal endoscopies as part of their normal medical care and deemed necessary by their physicians
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2043-02-28 (Estimated)

PRIMARY OUTCOMES:
Development of malignancy | Up to 20 years
  Assessment of participants for the development of malignancy during a 20-year follow-up period.

SECONDARY OUTCOMES:
Development of biomarkers | Up to 20 years
  To identify proteins, RNA and DNA that have changes in expression in those who develop cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Elham Afghani, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States